CLINICAL TRIAL: NCT07221214
Title: GLP-1 Receptor Agonists to Decrease Ethanol and CVD Risk in HIV - GL1DER HIV RCT
Brief Title: GLP-1 Receptor Agonists to Decrease Ethanol and CVD Risk in HIV
Acronym: GL1DER HIV RCT
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Norton Healthcare (Other); University of Louisville (Other)
Responsible Party: Principal Investigator, Hilary Tindle, Professor of Medicine, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1P60AA032176 (NIH); 1P60AA032176 (NIH)
Record Dates: First submitted 2025-10-23; First posted 2025-10-27 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: HIV; Alcohol; Smoking Cigarette; Cardiovascular Disease Prevention
Keywords: HIV; alcohol; smoking; tobacco; cardiovascular disease
MeSH Terms: conditions — Cigarette Smoking; Smoking; Cardiovascular Diseases | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Semaglutide (Experimental): drug intervention
  Interventions: Drug: Semaglutide (Rybelsus®)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide (Rybelsus®) — experimental study medication
  Arms: Semaglutide
Drug: Placebo — Placebo study product
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if the drug semaglutide works to reduce alcohol intake among adults living with HIV. The main questions it aims to answer are:

1. Does semaglutide lower the average number of alcoholic beverages participants drink per week?
2. Does semaglutide lower the average number of cigarettes participants smoke per day?
3. Does semaglutide decrease the risk for cardiovascular disease among people living with HIV who drink alcohol and/or smoke tobacco?

Researchers will compare the effects of semaglutide to a placebo (a look-alike substance that contains no drug) to see if semaglutide works to lower the alcohol intake among participants each week.

Participants will:

1. Take semaglutide for 3 months
2. Visit the research clinic 3 times for checkups and tests
3. Provide blood samples, stool samples, and saliva samples for tests.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18-89
* Prior diagnosis of HIV-1
* Affiliated with Vanderbilt Comprehensive Care Clinic
* On current ART regimen for at least 90 days prior to study entry with no missed doses for at least 7 consecutive days.
* Most recent absolute CD4 count ≥ 300 cells/mm3 and drawn within 12 months of study enrollment
* BMI ≥ 23 (calculated at screening)
* Self-report of consuming alcohol in past 90 days
* AUDIT-C ≥ 3 (male)/ ≥ 2 (female)
* Has an established stable address at which they can receive mail and can be reached for the next 6 months
* Willing and able to complete study procedures and follow-ups

Exclusion Criteria:

* Known allergy to semaglutide
* Currently taking GLP-1 RA (in the past 3 months)
* History of diabetes defined by diagnosis in Problems List in medical record
* History of pancreatitis
* History of gastroparesis
* Gallbladder disease (in the past 3 months)
* History of medullary thyroid carcinoma
* Family history of medullary thyroid carcinoma
* History of multiple endocrine neoplasia syndrome type 2
* Family history of multiple endocrine neoplasia syndrome type 2
* Cognitive inability to consent
* Barrier to speaking, hearing, reading, or writing English
* Pregnant or breastfeeding, or planning to become pregnant in the next 6 months
* Too ill to complete study procedures

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2026-02-06 (Estimated); Primary Completion 2029-07-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Average drinks/week past 30 days at 3 months | 3 Months
  Average drinks/week past 30 days (via Timeline Follow Back (TLFB))

SECONDARY OUTCOMES:
Average cigarettes per day (cpd) past 30 days at 3 months | 3 Months
  Average cigarettes per day in the past 30 days (via TLFB)
Systemic inflammation (IL-6) at 3 months | 6 Months
  Biomarker of systemic inflammation, Biomarker of gut permeability, Reynolds Risk Score, Mortality risk

CONTACTS AND LOCATIONS:
Overall Officials: Hilary A Tindle, MD, MPH, Principal Investigator — Vanderbilt University Medical Center

IPD SHARING:
Plan to Share IPD: No